CLINICAL TRIAL: NCT02087059
Title: A Multicenter, Open-label Clinical Study of the JAK Inhibitor Ruxolitinib (INC424) in Patients With Primary Myelofibrosis, Post-polycythemia Vera Myelofibrosis, or Post-essential Thrombocythemia Myelofibrosis
Brief Title: A Clinical Study of Ruxolitinib in Patients With Primary Myelofibrosis (PM), Post-polycythemia Vera (PV) Myelofibrosis, or Post-essential Thrombocythemia (ET) Myelofibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC424AJP01
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-05

CONDITIONS: Primary Myelofibrosis (MF)
Keywords: Post-Polycythemia Vera (PV) MF; Post-Essential Thrombocythemia (ET) MF
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ruxolitinib (Experimental): Ruxolitinib was administered orally twice daily at the starting dose of 5 mg, 15 mg or 20 mg bid based on Baseline platelet counts. The dosage was subsequently adjusted for safety and efficacy so that each patient was titrated to their most appropriate dose.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib

SUMMARY:
This is an open-label, multicenter clinical study in order to collect and examine data concerning the safety and efficacy of ruxolitinib in patients with Primary Myelofibrosis (MF), Post-Polycythemia Vera (PV) MF, Post-Essential Thrombocythemia (ET) MF.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Diagnosis of PMF, PPV-MF, or PET-MF, regardless of JAK2 mutational status. The diagnostic of PMF will be according to the World Health Organization (WHO) criteria (Thiele et al., 2008) and PPV-MF and PET-MF according to the International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) criteria (Barosi et al., 2008).
3. At least one risk factors provided in the definition of IWG-MRT (Cervantes et al., 2009; classified as intermediate risk-1, intermediate risk-2, or high risk)
4. Patients with intermediate risk-1 (patients who have only one of the IMG-MRT risk factors indicated above ) must have palpable splenomegaly with a length of ≥5 cm from the costal margin to the point of the greatest spleen protrusion.
5. Proportion of blasts in peripheral blood <10%
6. ECOG performance status of 0 to 2
7. The following values for bone marrow function prior to treatment:

   1. Absolute neutrophil count ≥1,000/μL, and
   2. Platelet count ≥50,000/μL without administration of a growth factor, thrombopoietin, or platelet transfusion
8. Stem cell transplantation is not a treatment option at present because it is not indicated or because there are no suitable donors.
9. All drugs used to treat MF were discontinued at least 28 days before treatment initiation.
10. Informed consent form should be signed before any screening procedures is performed

Exclusion Criteria:

1. Hepatic or renal impairment as indicated by the following:

   * Direct bilirubin ≥2-fold than the upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) >2.5-fold ULN
   * Creatinine >2.0 mg/dL
2. Clinically significant infection by bacteria, fungus, mycobacteria, parasite, or virus (screening and enrollment postponed until completion of antibiotic treatment in patients with an acute bacterial infection that requires antibiotic use)
3. Active hepatitis A, B, or C or HIV infection defined by a positive IgM-HA Ab test [hepatitis A virus antibody (immunoglobulin M [IgM])], HBs Ag test (hepatitis B surface antigen), HCV Ab test (hepatitis C virus antibody), or HIV Ab (human immunodeficiency virus antibody) at screening.
4. History of malignancy within the previous 3 years, except for early-stage squamous cell carcinoma and basal cell carcinoma.
5. History of serious congenital or acquired hemorrhagic disease
6. Previous platelet count <25,000/μL or absolute neutrophil count <500/μL, except for patients currently undergoing treatment for a myeloproliferative neoplasm or cytotoxic therapy for any other reason.
7. Splenic irradiation within 12 months before screening
8. Administration of hematopoietic growth factor receptor agonists (erythropoietin, granulocyte colony stimulating factor, romiplostim, eltrombopag) within 14 days before screening or 28 days before treatment initiation.
9. Currently receiving another investigational drug, or received another investigational drug within 30 days before the start of treatment.
10. History of myocardial infarction or acute coronary syndrome within 6 months before screening
11. Poorly controlled or unstable angina at present
12. Rapid or paroxysmal atrial fibrillation at present
13. Active alcohol or drug addiction that could hinder the patient's ability to comply with the study's requirements
14. Pregnant or currently breastfeeding woman
15. Women of childbearing potential or men with reproductive ability who are unwilling to take appropriate contraception measures
16. Patient with any concurrent condition that, in the Investigator's opinion, would jeopardize the safety of the patient or compliance with the protocol
17. History of hypersensitivity to the study drug or a drug with a similar chemical structure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- Japan (23):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Akita, Akita
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Tōon, Ehime
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Gifu, Gifu
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Miyazaki, Miyazaki
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Hirakata, Osaka
  - Novartis Investigative Site, Sayama, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Chūō, Yamanashi

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ruxolitinib
Started | 51
Completed | 44
Not Completed | 7
Not completed — Disease Progression | 1
Not completed — Adverse Event | 5
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Time Frame: 24 weeks
Measure: Number; unit: Participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 51
Participants
  AEs, regardless of study treatment relationship | 50
  AEs suspected to be related to study treatment | 46
  SAEs, regardless of study treatment relationship | 12
  SAEs suspected to be related to study treatment | 5
  AEs of CTC grade 3/4, regardless study treatment | 36
  AEs of CTC grade 3/4 suspected related treatment | 33
  AEs leading to the study treatment discontinuation | 5
  AEs requiring reduction or interruption treatment | 38
  AEs requiring concomitant medication | 33

2. Secondary Outcome: Charge in Spleen Size From Baseline at Specified Week
Description: Number of patients with spleen length reduced by ≥ 50% at specified week
Time Frame: Baseline, 24 weeks
Measure: Number; unit: particiapants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 51
particiapants
  Week 2 | 12
  Week 4 | 14
  Week 8 | 14
  Week 12 | 11
  Week 16 | 14
  Week 20 | 13
  Week 24 | 15

3. Secondary Outcome: Charge in Spleen Size From Baseline up to the Specified Week
Description: Number of patients with spleen length reduced by ≥ 50% up to specified week
Time Frame: Baseline, 24 weeks
Measure: Number; unit: particiapants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 51
particiapants
  Week 4 | 18 [13.1 to 38.2]
  Week 8 | 22 [16.2 to 42.5]
  Week 12 | 23 [16.2 to 42.5]
  Week 16 | 26
  Week 20 | 26
  Week 24 | 26

4. Secondary Outcome: Summary of Total Symptom Score as Measured by Seven-day Modified Myelofibrosis Symptom Assessment Form (MFSAF) v2.0 by Time
Description: The modified MFSAF v2.0 diary captures a patient's symptom severity on a scale of 0 (absent) to 10 (worst imaginable),with a maximal summary score of 60
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 51
score on a scale
  Night Sweats baseline (n=51) | 2.9 (3.07)
  Night Sweats week 24 (n=43) | 0.6 (1.35)
  Itching baseline (n=51) | 1.8 (2.39)
  Itching week 24 (n=43 | 0.6 (1.25)
  Abdominal Discomfort baseline( n=51) | 4.4 (3.18)
  Abdominal Discomfort week 24(n=43) | 1.4 (1.84)
  Pain under ribs on left Baseline (=51) | 2.2 (2.72)
  Pain under ribs on left week 24 (=43) | 0.7 (1.26)
  Feeling of fullness Baseline (n=51) | 3.2 (2.91)
  Feeling of fullness week 24 (n=43) | 1.3 (1.8)
  Bone/muscle pain Baseline (n=51) | 2.3 (2.83)
  Bone/muscle pain week 24 (n=43) | 1.0 (1.83)
  Degree of inactivity Baseline (n=51) | 2.3 (2.84)
  Degree of inactivity week 24 (n=43) | 1.0 (1.66)
  Total symptom score baseline (n=51) | 16.8 (12.30)
  Total symptom score week 24 (n=43) | 5.7 (6.48)

5. Secondary Outcome: Summary of Summary of EORTC QLQ-C30 Responses by Time
Description: The QLQ-C30 version 1.0 (QLQ-C30) incorporates five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health status / QoL scale, and a number of single items assessing additional symptoms commonly reported by cancer patients (dyspnoea, loss of appetite, insomnia, constipation and diarrhea) and perceived financial impact of the disease.All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Time Frame: 24 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 51
units on a scale
  Physical Functioning baseline | 79.35 (17.951)
  Physical Functioning 24(n=43) | 86.67 (17.959)
  Role Functioning Baseline(n=51) | 77.78 (23.254)
  Role Functioning Week 24(n=43) | 83.72 (19.068)
  Emotional Functioning Baseline(n=51) | 85.46 (17.705)
  Emotional Functioning Week 24(n=43) | 92.05 (13.357)
  Cognitive Functioning Baseline(n=51) | 78.43 (20.356)
  Cognitive Functioning week 24 (n=43) | 79.84 (17.653)
  Social Functioning Baseline (n=51) | 85.62 (19.154)
  Social Functioning week 24(n=43) | 87.60 (17.852)
  Global Health Status/QOL Baseline (n=51) | 55.72 (22.882)
  Global Health Status/QOL week 24 (n=43) | 66.47 (22.456)
  Fatigue Baseline(n=51) | 40.31 (23.787)
  Fatigue week 24 (n=43) | 28.68 (23.412)
  Nausea and Vomiting baseline (n=51) | 4.90 (13.862)
  Nausea and Vomiting week 24 (n=43) | 0.39 (2.542)
  Pain Baseline | 21.57 (21.678)
  Pain week 24 (n=43) | 10.08 (15.911)
  Dyspnoea baseline (n=51) | 22.88 (25.377)
  Dyspnoea Week 24 (n=43) | 25.58 (23.946)
  Insomnia baseline (n=51) | 23.53 (29.283)
  Insomnia Week 24 (n=43) | 15.50 (23.400)
  Appetite Lose baseline (n=51) | 21.57 (27.787)
  Appetite Lose Week 24 (n=43) | 9.30 (16.786)
  Constipation baseline (n=51) | 8.50 (20.916)
  Constipation Week 24 (n=43) | 8.53 (16.416)
  Diarrhoea baseline (n=51) | 18.30 (24.325)
  Diarrhoea Week 24 (n=43) | 12.40 (23.029)
  Financial Difficulties baseline (n=51) | 15.69 (25.257)
  Financial Difficulties Week 24 (n=43) | 20.93 (30.012)

ADVERSE EVENTS:
Arm/Group | Ruxolitinib
Serious Adverse Events (participants affected / at risk) | 12/51
Other Adverse Events (participants affected / at risk) | 49/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=51)
Anaemia (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Multi-organ failure (General disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Empyema (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Gout (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Withdrawal syndrome (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=51)
Anaemia (Blood and lymphatic system disorders) | 32
Leukopenia (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 15
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 5
Hepatic function abnormal (Hepatobiliary disorders) | 6
Nasopharyngitis (Infections and infestations) | 6
Pneumonia (Infections and infestations) | 4
Electrocardiogram QT prolonged (Investigations) | 5
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 12
Weight increased (Investigations) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary.

However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.